CLINICAL TRIAL: NCT05377762
Title: Validation of an Italian Questionnaire of Adherence to the Ketogenic Diet: iKetoCheck
Brief Title: Validation of an Italian Questionnaire of Adherence to the Ketogenic Diet
Acronym: iKETOCHECK
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Pavia (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor
Other Study IDs: iKETOCHECK
Record Dates: First submitted 2022-05-10; First posted 2022-05-17 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-05

CONDITIONS: Epilepsy
Keywords: ketogenic diet; adherence; questonnaire
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ketogenic diet (KD) represents an effective and safe non-drug treatment for drug-resistant epilepsy in pediatric and adult age based on normocaloric, hyperlipidic (80-90% of the daily energy), normoproteic and hypoglucidic dietary regimen. Adherence to treatment with KD is often difficult in the long term, for the patient and for caregivers, especially in adolescence. There are no tools in the literature other than monitoring ketonemia to measure adherence to the diet. A quality tool, validated by experts, on a large population, would allow for a more solid assessment of adherence to treatment, facilitating clinicians in the interpretation of efficacy results and in implementing an early intervention to adjust the therapy.

DETAILED DESCRIPTION:
The ketogenic diet (KD) represents an effective and safe non-drug treatment for drug-resistant epilepsy in pediatric and adult age and is the gold standard therapy for type I glucose transporter deficiency syndrome (GLUT1 DS). According to international guidelines, once undertaken, the KD must be continued for at least three months in order to determine its effectiveness and can be continued for years if effective.

In summary, KD is a normocaloric, hyperlipidic (80-90% of the daily energy), normoproteic and hypoglucidic dietary regimen that determines in the organism a state of ketosis similar to that induced by a prolonged fast, which corresponds to average levels of ketonemia equal to 2.5 mmol / L.

Not being able to estimate the concentration of ketone bodies in the brain, the serum measurement is adopted, i.e. the detection of capillary ketonemia. It is important to consider the presence of inter-individual and intra-individual variability of ketonemia and this can be influenced by various factors in addition to the composition of the diet and the ketogenic ratio (fat / protein + carbohydrates): infectious episodes, physical activity, hydration , steroid therapy. Hence the importance of individualized treatment and careful monitoring of adherence to dietary recommendations. The quality of the diet, especially at the beginning of ketogenic therapy, but during the entire follow-up, is essential for achieving optimal levels of ketosis.However, adherence to treatment with KD is often difficult in the long term, for the patient and for caregivers, especially in adolescence. Failure to adhere to KD is mainly attributed to dietary side effects, psychosocial factors, or the dietary restriction itself.

There are no tools in the literature other than monitoring ketonemia to measure adherence to the diet; usually, clinicians ask parents and patients to share the food diary in order to check the calorie intake, the ketogenic ratio and the nutritional composition of the diet. A 'Keto-check' questionnaire was recently developed and validated in Brazil, currently only available in Portuguese, with the aim of providing a tool to measure adherence to the ketogenic diet through simple, easily reproducible questions. A quality tool, validated by experts, on a large population, would allow for a more solid assessment of adherence to treatment, facilitating clinicians in the interpretation of efficacy results and in implementing an early intervention to adjust the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age <60 years
* Gender: both sexes
* Route of administration of the diet: totally or partially oral
* Diagnosis: drug-resistant epilepsy or GLUT1 deficiency
* Duration of treatment with the ketogenic diet: at least 3 months
* Informed consent of the patient and / or an authorized caregiver / legal representative•

Exclusion Criteria:

* Age > 60 years
* Route of administration of the exclusively enteral or parenteral diet
* Duration of treatment with KD less than 3 months

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients treated with a ketogenic diet for more than three months belonging to the Center for Childhood and Adolescent Epileptology of the Mondino Foundation of Pavia will be enrolled, who will accept to participate in the study and will have signed the relative informed consent. For patients under the age of 18, the answers to the questionnaire and the related informed consent must be provided by the parents or legal guardian.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Adherence score | Through study completion, an average of 6 months
  The answer of questionnaire will generate a score. Minimum value will be 10 points and maximum 50 points. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Valentina De Giorgis, Principal Investigator — University of Pavia
Locations (2):
- Italy (2):
  - University of Pavia, Pavia
  - Center for Childhood and Adolescent Epileptology of the Mondino Foundation, Pavia

IPD SHARING:
Plan to Share IPD: Undecided